CLINICAL TRIAL: NCT05374252
Title: A Phase 3, Multicenter, Double-Blind Randomized Study of Mitomycin, 5-Fluorouracil and IMRT Combined With or Without Anti-PD-1 in Patients With Locally Advanced Anal Canal Squamous Carcinoma
Brief Title: Chemoradiotherapy Combined With or Without PD-1 Blockade in Anal Canal Squamous Carcinoma Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2021144
Record Dates: First submitted 2022-05-10; First posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Anal Canal Cancer Stage III; Anal Squamous Cell Carcinoma; Anal Canal Cancer; Anal Cancer
Keywords: Anal Squamous Cell Carcinoma; Radiochemotherapy; PD-1
MeSH Terms: conditions — Anal Canal Carcinoma; Anus Neoplasms | interventions — Immune Checkpoint Inhibitors; Radiation; Chemoradiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): Concurrent PD-1 antibody sintilimab combined with mytomicin C, 5-fluorouracil, and IMRT, followed by adjuvant sintilimab
  Interventions: Drug: PD-1 inhibitor
- Control Group (Active Comparator): Concurrent mytomicin C and 5-fluorouracil combined with IMRT
  Interventions: Radiation: concurrent chemoradiotherapy

INTERVENTIONS:
Drug: PD-1 inhibitor — Two cycles of concurrent PD-1 antibody sintilimab combined with mytomicin C, 5-fluorouracil and IMRT, followed by adjuvant sintilimab for six months
  Other Names: radiation; concurrent chemotherapy
  Arms: Experimental Group
Radiation: concurrent chemoradiotherapy — Two cycles of concurrent mytomicin C and 5-fluorouracil combined with IMRT
  Other Names: radiation; concurrent chemotherapy
  Arms: Control Group

SUMMARY:
This is a phase III, multi-center, double-blind randomized controlled trial assessing the efficacy and safety of concurrent mitomycin C/5-Fu chemotherapy and long-course IMRT combined with PD-1 antibody Sintilimab for locally advanced anal canal squamous carcinoma patients, by comparing an experiment group (traditional chemoradiotherapy with PD-1 antibody Sintilimab) with a control group (traditional treatment without Sintilimab).

ELIGIBILITY:
Inclusion Criteria:

1. Histology identified anal canal squamous carcinoma,
2. Aged 18 to 75,
3. Clinical staging III, Eastern Cooperative Oncology Group 0-2 score,
4. The Staging method: All patients undergoing rectal anus palpation, high resolution MRI and chest-abdominal enhanced CT, clinical data should be re-evaluated and inclusive by center evaluation group when there is contradictory staging, distant metastasis were excluded by chest-abdominal enhanced CT and pelvic enhanced MRI,
5. No previous anal canal surgery or anal tumor resection (except for biopsy),
6. No previous chemotherapy or pelvic radiotherapy history,
7. No biopharmaceutical treatment history (such as monoclonal antibody), immunotherapy (such as anti PD-1antibody, anti PD-L1 antibody, anti PD-L2 antibody or anti CTLA-4), or other research drug treatment in the previous 5 years,
8. Adequate bone marrow, liver, and kidney function,
9. Clinical complete response (cCR) (Chest, abdominal and pelvic enhanced CT or pelvic enhanced MRI or PET/CT),
10. Informed consent assigned, Final inclusion criteria,
11. Non-pregnant or breast-feeding women,
12. No other malignant disease within 5 years before diagnosis of anal cancer squamous carcinoma (except endocervical cancer in situ or skin basal cell carcinoma which had been cured); no other malignant disease beside anal cancer squamous carcinoma,
13. No other serious disease leading to shortened survival.

Exclusion Criteria:

1. Diagnosed as stage I-II and well differentiated squamous cell carcinoma,
2. Distant metastasis,
3. Received radiation therapy in abdominal or pelvic regions,
4. Pregnant, lactating woman patient or fertile but lacks adequate contraceptives,
5. Arrhythmia need anti-arrhythmia treatment (except β-blocking agent or Digoxin), symptomatic coronary heart disease or myocardial ischemia (myocardial infarction within 6 months) or congestive heart-failure (CHF) > New York Heart Association grade II,
6. Severe hypertension not well controlled by drugs,
7. Active phase of chronic hepatitis B or hepatitis C (high copies of virus DNA),
8. Patients with active tuberculosis (TB) are receiving anti-tuberculosis treatment or have received anti-tuberculosis treatment within 1 year before screening,
9. Other active clinical severe infection (NCI-CTCAE (version 4.0) ),
10. Dyscrasia, organ dysfunction,
11. Known or suspicious allergy to any research-related drugs,
12. Epilepsy needs treatments (Steroid or anti-epilepsy therapy),
13. Other malignant tumor history within 5 years,
14. Drug abuse and medical, psychological, or social factors that may interfere with patients' participation in the study or affect the evaluation of the study,
15. Patients have any active autoimmune diseases or a history of autoimmune diseases (including but not restricted: interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, nephritis, hyperthyroidism and decreased thyroid function; patients with vitiligo or with complete remission of asthma in childhood and without any intervention in adulthood may be included; patients with asthma requiring bronchodilators intervention are not included,
16. Any anti-infection vaccine 4 weeks before inclusion,
17. Long-term exposure to immune-suppressor, combination of systemic or topical use of corticosteroids (dose>10mg/day prednisolone or equivalent hormone),
18. Any unstable state might endanger the patients' safety and compliance,
19. Refuses to sign informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2022-05-07 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | from the end of treatment to 3 years after treatment
  progression free survival
Overall survival | from the end of treatment to 3 years after treatment
  overall survival
cCR rate | 6 months after treatment
  cCR rate 6 months after treatment

SECONDARY OUTCOMES:
Acute toxicities | from the start of treatment to 3 months after treatment
  acute toxicities according to the NCI CTCAE (version 4.0)
cCR rate | 3 months after treatment
  cCR rate 3 months after treatment
The rate of late toxicity according to the RTOG/EORTC scale | 3 years
  The rate of late toxicity according to the RTOG/EORTC scale
Colostomy rate | 2 year
  colostomy rate
Local recurrence rate | from the end of treatment to 3 years after treatment
  local recurrence rate
Distant metastasis rate | from the end of treatment to 3 years after treatment
  distant metastasis rate
Incidence rate of Grade ≥3 PD-1monoclonal antibody-related adverse events | 1 year
  Incidence rate of Grade ≥3 PD-1monoclonal antibody-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Xiang-bo Wan, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Bartelink H, Roelofsen F, Eschwege F, Rougier P, Bosset JF, Gonzalez DG, Peiffert D, van Glabbeke M, Pierart M. Concomitant radiotherapy and chemotherapy is superior to radiotherapy alone in the treatment of locally advanced anal cancer: results of a phase III randomized trial of the European Organization for Research and Treatment of Cancer Radiotherapy and Gastrointestinal Cooperative Groups. J Clin Oncol. 1997 May;15(5):2040-9. doi: 10.1200/JCO.1997.15.5.2040. PMID 9164216
- [Result] Gunderson LL, Moughan J, Ajani JA, Pedersen JE, Winter KA, Benson AB 3rd, Thomas CR Jr, Mayer RJ, Haddock MG, Rich TA, Willett CG. Anal carcinoma: impact of TN category of disease on survival, disease relapse, and colostomy failure in US Gastrointestinal Intergroup RTOG 98-11 phase 3 trial. Int J Radiat Oncol Biol Phys. 2013 Nov 15;87(4):638-45. doi: 10.1016/j.ijrobp.2013.07.035. Epub 2013 Sep 10. PMID 24035327
- [Result] James RD, Glynne-Jones R, Meadows HM, Cunningham D, Myint AS, Saunders MP, Maughan T, McDonald A, Essapen S, Leslie M, Falk S, Wilson C, Gollins S, Begum R, Ledermann J, Kadalayil L, Sebag-Montefiore D. Mitomycin or cisplatin chemoradiation with or without maintenance chemotherapy for treatment of squamous-cell carcinoma of the anus (ACT II): a randomised, phase 3, open-label, 2 x 2 factorial trial. Lancet Oncol. 2013 May;14(6):516-24. doi: 10.1016/S1470-2045(13)70086-X. Epub 2013 Apr 9. PMID 23578724
- [Result] Ben-Josef E, Moughan J, Ajani JA, Flam M, Gunderson L, Pollock J, Myerson R, Anne R, Rosenthal SA, Willett C. Impact of overall treatment time on survival and local control in patients with anal cancer: a pooled data analysis of Radiation Therapy Oncology Group trials 87-04 and 98-11. J Clin Oncol. 2010 Dec 1;28(34):5061-6. doi: 10.1200/JCO.2010.29.1351. Epub 2010 Oct 18. PMID 20956625
- [Result] Ott PA, Piha-Paul SA, Munster P, Pishvaian MJ, van Brummelen EMJ, Cohen RB, Gomez-Roca C, Ejadi S, Stein M, Chan E, Simonelli M, Morosky A, Saraf S, Emancipator K, Koshiji M, Bennouna J. Safety and antitumor activity of the anti-PD-1 antibody pembrolizumab in patients with recurrent carcinoma of the anal canal. Ann Oncol. 2017 May 1;28(5):1036-1041. doi: 10.1093/annonc/mdx029. PMID 28453692
- [Result] Shahjehan F, Kamatham S, Ritter A, Kasi PM. Dramatic response to modified docetaxel, cisplatin, and fluorouracil chemotherapy after immunotherapy in a patient with refractory metastatic anal cancer. Clin Case Rep. 2019 Aug 6;7(9):1729-1734. doi: 10.1002/ccr3.2333. eCollection 2019 Sep. PMID 31534737
- [Result] Nigro ND, Vaitkevicius VK, Considine B Jr. Combined therapy for cancer of the anal canal: a preliminary report. Dis Colon Rectum. 1974 May-Jun;17(3):354-6. doi: 10.1007/BF02586980. No abstract available. PMID 4830803
- [Result] Northover J, Glynne-Jones R, Sebag-Montefiore D, James R, Meadows H, Wan S, Jitlal M, Ledermann J. Chemoradiation for the treatment of epidermoid anal cancer: 13-year follow-up of the first randomised UKCCCR Anal Cancer Trial (ACT I). Br J Cancer. 2010 Mar 30;102(7):1123-8. doi: 10.1038/sj.bjc.6605605. Epub 2010 Mar 16. PMID 20354531
- [Result] Epidermoid anal cancer: results from the UKCCCR randomised trial of radiotherapy alone versus radiotherapy, 5-fluorouracil, and mitomycin. UKCCCR Anal Cancer Trial Working Party. UK Co-ordinating Committee on Cancer Research. Lancet. 1996 Oct 19;348(9034):1049-54. PMID 8874455